CLINICAL TRIAL: NCT01637324
Title: The Thai Red Cross AIDS Research Centre
Brief Title: Multidisciplinary Services to Enhance HIV Testing and Linkage to Care Among MSM
Status: Completed | Type: Observational
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Collaborators: National Institutes of Health (NIH) (NIH); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MSM VCT
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: HIV Testing; Linkage to Care
Keywords: To assess VCT and linkage into care; nPEP; STIs; anal dysplasia/cancer; hyperlipidemia; diabetes; Proportion of first-time MSM clients attending multidisciplinary services who undergo HIV testing; Proportion of MSM clients who have repeated HIV testing during the first six months after the first negative HIV test; Proportion of HIV-positive MSM who receive HIV care within three months after HIV diagnosis or enrolment; Proportion of HIV-positive MSM who still remain in HIV care at six months after enrollment
MeSH Terms: conditions — Sexually Transmitted Diseases; Neoplasms; Hyperlipidemias; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives

1. To determine the impact of MSM-targeted multidisciplinary services on uptake of HIV voluntary counseling and testing (VCT)
2. To determine the impact of MSM-targeted multidisciplinary services on the enrollment into care and retention of HIV-positive MSM

Subject population: HIV-negative and HIV-positive MSM clients, age ≥18 years old, of the Thai Red Cross Anonymous Clinic (TRC-AC) in Bangkok Thailand, the Cipto Mangunkusumo Hospital in Jakarta, and the Sanglah Hospital in Bali, Indonesia

Number of participants: 200 HIV-negative and 150 HIV-positive MSM participants

DETAILED DESCRIPTION:
This is a prospective cohort study which will recruit 350 MSM clients within 3 months, and follow them for 12 months. MSM to be recruited will be first-time clients who come to the clinics for services other than VCT. These services may include but would not be limited to sexually transmitted infection (STI) diagnosis and treatment, anal dysplasia screening, nutritional counseling and non-occupational post-exposure prophylaxis (nPEP).

Approximately 250 MSM clients with unknown or previously negative HIV status will be offered HIV testing every 3 months (HIV-negative MSM cohort). MSM from the HIV-negative cohort who tested HIV-positive during the study (estimated 20%, 50 MSM) will be referred to the HIV-positive MSM cohort and will be followed up every 6 months. Additional clients who visit the clinic during the 3-month recruitment period with previously known HIV-positive status but have not been linked to HIV care (up to 100) will also be enrolled into HIV-positive MSM cohort. Therefore, there will be up to 150 HIV-positive subjects enrolled in this study. Each enrolled participant will have 12 months in the study.

This study will allow us to assess VCT and linkage into care, as well as HIV risk behavior and need for nPEP, and the incidence or prevalence of important morbidities in MSM such as STIs, anal dysplasia/cancer, hyperlipidemia, and diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male with history of anal sex with men
2. Age 18 years old or older
3. Thai or Indonesian citizen as identified by the Thai or Indonesian National Identification card
4. Willing to provide location or contact information and allow contact
5. Live in or near Bangkok, Jakarta, or Bali and is available for follow-up for the planned study duration
6. Understand the study and sign informed consent form.

Exclusion Criteria:

1. Persons who have a history of a medical or psychiatric disorder by investigator's interview and physical examination according to standard practices, that in the judgment of the investigator(s), would interfere with ability to give informed consent.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSM with HIV negative and positive MSM in Thai Red Cross Bangkok Thailand, the Cipto Mangunkusumo Hospital in Jakarta, and the Sanglah Hospital in Bali, Indonesia
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Thai Red Cross AIDS Research Centre, Pathumwan, Bangkok, Thailand